CLINICAL TRIAL: NCT04009304
Title: Effective Training Models for Implementing Health-Promoting Practices Afterschool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Rebekka Lee, Research Scientist, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6928483
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Obesity, Childhood
Keywords: Nutrition; Physical activity
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Assigned afterschool sites (not individual participants) to group with block randomization approach, delayed intervention design offered effective intervention to control group in year 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-person (Experimental): OSNAP intervention delivered to afterschool sites using an in-person train-the-trainer model implementation strategy
  Interventions: Behavioral: OSNAP
- Online (Experimental): OSNAP intervention delivered to afterschool sites using an online training model implementation strategy
  Interventions: Behavioral: OSNAP
- Control (No Intervention)

INTERVENTIONS:
Behavioral: OSNAP — Afterschool practice and policy change to support healthy eating and physical activity
  Arms: In-person; Online

SUMMARY:
This study of the dissemination of the Out-of-school Nutrition and Physical Activity Initiative will utilize a 3-arm group-randomized control trial to establish the effectiveness of two learning collaborative training models (e.g. train-the-trainer in-person vs. online) for an evidence-based out-of-school time (OST) nutrition and physical activity intervention. The study will compare sites that receive the training models with a control group. Investigators will work with YMCA leadership to recruit 45 demographically diverse YMCA OST sites from across the country. Sites will be matched on racial/ethnic composition, proportion of students eligible for free or reduced price meals, program enrollment, urban/rural/suburban setting, and physical activity and food service facilities available. One-third of the sites will be randomized to participate in the online training over the school year, one-third will participate in the in-person train-the-trainer model, and one-third will serve as controls. After randomization, in fall 2016, teams of YMCA OST directors and line staff will be invited to participate in the OSNAP learning collaborative trainings. The intervention follows the social ecological model with activities targeting multiple levels of change-school district/program sponsor, OST site, interpersonal, and individual-and emphasizing on adoption of the following OSNAP goals: ban sugar-sweetened drinks from snacks served and brought in from outside the snack program; offer water as a drink at snack every day; offer a fruit or vegetable option every day at snack; ban foods with trans fats from snacks served; serve whole grains; offer 30 minutes of physical activity to all children daily; offer 20 minutes of vigorous physical activity to all children 3 times per week; and eliminate television, movies, and non-educational screentime. Sessions are designed consistent with the Institute for Healthcare Improvement Breakthrough Series Collaborative model and use constructs from social cognitive theory-knowledge and skill development coupled with action planning-to drive environmental and behavior change. Teams of afterschool staff will use the Out-of-School Nutrition and Physical Activity Observational Practice Assessment Tool (OSNAP-OPAT), decision aids, policy writing guides, and other resources available at www.osnap.org to set data-driven goals and implement discrete practice, policy, and communication action steps throughout the year. Staff will also receive training on the Food & Fun After School curriculum available at foodandfun.org.

ELIGIBILITY:
Inclusion Criteria:

* Staff from afterschool sites that are run by the YMCA
* Staff from afterschool sites that serve elementary age children
* Staff from afterschool sites that run programming for the duration of the school year

Exclusion Criteria:

- Staff from afterschool sites that have already had experience implementing the OSNAP intervention

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in nutrition and physical activity goals met (aggregate score) | Measured pre/post about 6 months apart
  Effectiveness of the intervention will be measured with the Out-of-School Nutrition and Physical Activity Observational Practice Assessment Tool (OSNAP-OPAT)-an observational measure of nutrition and physical activity practices that site staff complete for one week before and after the intervention. Our team validated the tool with OST staff similar to those proposed to complete the measure in this study, establishing criterion validity for physical activity and nutrition outcomes with correlations ranging from 0.56 to 0.85 when compared with accelerometry and direct observation of dietary intake.
  Minimum goals possible: 0; Maximum goals possible: 9 Higher values represent better outcomes

SECONDARY OUTCOMES:
Change from baseline in % of days offering physical activity, screentime, fruits and vegetables, water, juice, whole grains, and sugary drinks from outside the program | Measured pre/post about 6 months apart
  Using same Out-of-School Nutrition and Physical Activity Observational Practice Assessment Tool (OSNAP-OPAT measure) - components of aggregate score Minimum days possible: 0%; Maximum days possible: 100% Higher values represent better outcomes

OTHER OUTCOMES:
Cost of the implementation strategy | Measured up to 1 year after baseline
  Data on personnel, travel, and material costs collected via activity logs and administrative records
Reach: number of children and afterschool staff impacted by each implementation strategy | Measured at baseline
  Collected on registration forms and via administrative records

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee RM, Barrett JL, Daly JG, Mozaffarian RS, Giles CM, Cradock AL, Gortmaker SL. Assessing the effectiveness of training models for national scale-up of an evidence-based nutrition and physical activity intervention: a group randomized trial. BMC Public Health. 2019 Nov 28;19(1):1587. doi: 10.1186/s12889-019-7902-y. PMID 31779603